CLINICAL TRIAL: NCT05952700
Title: Evaluation and Optimization of Machine Learning Algorithms for Individual Bladder Filling Level Prediction by a Sensor System
Brief Title: inContAlert: Machine Learning Algorithms for Individual Bladder Filling Level Prediction
Status: Completed | Type: Observational
Sponsor: inContAlert GmbH (Industry)
Collaborators: University of Bayreuth (Other)
Responsible Party: Sponsor
Other Study IDs: Az. O 1305/1 -GB
Record Dates: First submitted 2023-06-05; First posted 2023-07-19 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Monitoring of the Bladder Filling
Keywords: bladder monitoring; digital Health; bladder filling level; incontinence; neurourology; neurogenic bladder; spinal cord injury
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: inContAlert — InContAlert is a non-invasive sensor technology to measure the bladder filling level for incontinence patients. The device is fixed about 2cm above the pubic bone using a patch or strap and does not require surgery. The data collected from the patient is analyzed using deep learning algorithms. The bladder filling level determined in this way is then displayed on an app.

SUMMARY:
The aim of this study is to evaluate the bladder filling level of the study participants using the inContAlert sensor. The generated data will be used for the evaluation and optimization of the machine learning algorithms to be able to make precise predictions about the individual bladder fill level.

In particular, the hypothesis that the bladder filling level can be estimated by the algorithm will be tested. When testing the hypothesis, it should be determined which deviation (measured by the mean absolute percentage error) of the estimation/prediction differs from the actual value (obtained by measuring the urine output using a measuring cup in combination with kitchen scales).

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

* Missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The selection of the study participants is based on a voluntary basis by inContAlert GmbH.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Difference between the predicted bladder filling level and the actual value | December 2023
  Difference (measured as mean absolute error in percent) of the predicted bladder filling level (measured in ml) and the actual value (determined by measuring the volume of urine in ml with a measuring cup in combination with a kitchen scale).

CONTACTS AND LOCATIONS:
Overall Officials: Jannik Lockl, Dr., Study Director — inContAlert GmbH
Locations (1):
- inContAlert GmbH, Bayreuth, Germany

IPD SHARING:
Plan to Share IPD: No